CLINICAL TRIAL: NCT03519698
Title: Efficacy of Footbaths With Ginger, Mustard & Warm Water Only on Psychophysiological Parameters in Female Adolescents With & Without Anorexia Nervosa - a Randomized, Controlled, Three-arm Study With Cross-over Design
Brief Title: Footbaths With Ginger, Mustard & Warm Water Only in Female Adolescents With & Without Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Responsible Party: Principal Investigator, Dr. Jan Vagedes, Director, Clinical Research, ARCIM Institute Academic Research in Complementary and Integrative Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SWI_05
Record Dates: First submitted 2018-01-12; First posted 2018-05-09 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Amines; ginger extract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Warm water (Placebo Comparator): 12 l footbath with warm water (40 °C)
  Interventions: Other: Warm water
- Warm water & Mustard (Experimental): 12 l footbath with warm water (40 °C) and 80 g mustard flour
  Interventions: Other: Warm water; Other: Mustard
- Warm water & Ginger (Experimental): 12 l footbath with warm water (40 °C) and 80 g ginger flour
  Interventions: Other: Warm water; Other: Ginger

INTERVENTIONS:
Other: Warm water — Footbaths were prepared with 12 liters of warm water (40 °C)
Other: Mustard — 12 l footbath with warm water (40 °C) and 80 g mustard flour (Sinapis nigrea semen plv.)
  Other Names: Sinapis nigrea semen
  Arms: Warm water & Mustard
Other: Ginger — 12 l footbath with warm water (40 °C) and 80 g ginger flour (Zingiberis rhizoma plv.)
  Other Names: Zingiberis rhizoma
  Arms: Warm water & Ginger

SUMMARY:
A randomized, controlled, three-arm study to investigate the effects of footbaths with ginger, mustard or warm water alone in female, adolescent patients with Anorexia nervosa and in healthy, female adolescents on psychophysiological parameters.

DETAILED DESCRIPTION:
In a cross-over study design, the subjects (21 female patients with Anorexia nervosa, 20 healthy, female controls) receive footbaths with either ginger, mustard or warm water alone in a randomized order with a wash-out period of at least 1-3 days. The effects of each intervention on the objective warmth generation are measured by infrared thermography, whereas the subjective warmth perception is determined by the 'Herdecke warmth perception questionnaire'. All parameters are determined at specified times (t1 = right before, t2 = right after and t3 = 10 minutes following the footbath), which enables an evaluation based on pre-post-comparisons. The statistical analysis comprises analyses of variances based on linear mixed effects models (after checking for carry-over effects).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent of the parents
* Age 12-18 years

Exclusion Criteria:

* Infectious disease with body temperature above 38 °C
* Skin damages at the lower legs/feet
* Known intolerance/ anaphylaxis to mustard or ginger preparations
* Cardiac arrhythmia
* Pregnancy
* Insufficient knowledge of the German language
* BMI percentile < 10% (for control group)

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
Change in 2-Item Warmth Perception Measure (feet) from t1 to t3 | right before the footbath (t1) and 10 minutes following the footbath (t3)
  Self-reported warmth perception at both feet assessed with the "Herdecke warmth perception questionnaire" right before (t1) and 10 minutes following the footbath (t3). Each item is scored 0-4 (0 = cold; 4 = hot), yielding a total between 0 - 8.

SECONDARY OUTCOMES:
Change in 2-Item Warmth Perception Measure (feet) from t1 to t2 | right before the footbath (t1) and right after the footbath (t2, 5-20 minutes after t1 depending on the actual footbath length)
  Self-reported warmth perception at both feet assessed with the "Herdecke warmth perception questionnaire" right before (t1) and right after the footbath (t2). Each item is scored 0-4 (0 = cold; 4 = hot), yielding a total between 0 - 8.
Change in 2-Item Warmth Perception Measure (face) from t1 to t3 | right before the footbath (t1) and 10 minutes following the footbath (t3)
  Self-reported warmth perception in the face assessed with the "Herdecke warmth perception questionnaire" right before (t1) and 10 minutes following the footbath (t3). Each item is scored 0-4 (0 = cold; 4 = hot), yielding a total between 0 - 8.
Change in 2-Item Warmth Perception Measure (face) from t1 to t2 | right before the footbath (t1) and right after the footbath (t2, 5-20 minutes after t1 depending on the actual footbath length)
  Self-reported warmth perception in the face assessed with the "Herdecke warmth perception questionnaire" right before (t1) and right after the footbath (t2). Each item is scored 0-4 (0 = cold; 4 = hot), yielding a total between 0 - 8.
Change in 2-Item Warmth Perception Measure (hands) from t1 to t3 | right before the footbath (t1) and 10 minutes following the footbath (t3)
  Self-reported warmth perception at both hands assessed with the "Herdecke warmth perception questionnaire" right before (t1) and 10 minutes following the footbath (t3). Each item is scored 0-4 (0 = cold; 4 = hot), yielding a total between 0 - 8.
Change in 2-Item Warmth Perception Measure (hands) from t1 to t2 | right before the footbath (t1) and right after the footbath (t2, 5-20 minutes after t1 depending on the actual footbath length)
  Self-reported warmth perception at both hands assessed with the "Herdecke warmth perception questionnaire" right before (t1) and right after the footbath (t2). Each item is scored 0-4 (0 = cold; 4 = hot), yielding a total between 0 - 8.
Change in 1-Item Warmth Perception Measure (overall warmth) from t1 to t3 | right before the footbath (t1) and 10 minutes following the footbath (t3)
  Self-reported overall warmth perception assessed with the "Herdecke warmth perception questionnaire" right before (t1) and 10 minutes following the footbath (t3). The item is scored 0-4 (0 = cold; 4 = hot), yielding a total between 0 - 4.
Change in 1-Item Warmth Perception Measure (overall warmth) from t1 to t2 | right before the footbath (t1) and right after the footbath (t2, 5-20 minutes after t1 depending on the actual footbath length)
  Self-reported overall warmth perception assessed with the "Herdecke warmth perception questionnaire" right before (t1) and right after the footbath (t2). The item is scored 0-4 (0 = cold; 4 = hot), yielding a total between 0 - 4.
Change in Distal Skin Temperature Measure (feet) from t1 to t3 | right before the footbath (t1) and 10 minutes following the footbath (t3)
  Distal skin temperature in °C at both feet measured with a high-definition infrared camera (FLIR-Systems, type SC660) right before (t1) and 10 minutes following the footbath (t3).
Change in Distal Skin Temperature Measure (feet) from t1 to t2 | right before the footbath (t1) and right after the footbath (t2, 5-20 minutes after t1 depending on the actual footbath length)
  Distal skin temperature in °C at both feet measured with a high-definition infrared camera (FLIR-Systems, type SC660) right before (t1) and right after the footbath (t2).
Change in Distal Skin Temperature Measure (face) from t1 to t3 | right before the footbath (t1) and 10 minutes following the footbath (t3)
  Distal skin temperature in °C in the face measured with a high-definition infrared camera (FLIR-Systems, type SC660) right before (t1) and 10 minutes following the footbath (t3).
Change in Distal Skin Temperature Measure (face) from t1 to t2 | right before the footbath (t1) and right after the footbath (t2, 5-20 minutes after t1 depending on the actual footbath length)
  Distal skin temperature in °C in the face measured with a high-definition infrared camera (FLIR-Systems, type SC660) right before (t1) and right after the footbath (t2).
Change in Distal Skin Temperature Measure (hands) from t1 to t3 | right before the footbath (t1) and 10 minutes following the footbath (t3)
  Distal skin temperature in °C at both hands measured with a high-definition infrared camera (FLIR-Systems, type SC660) right before (t1) and 10 minutes following the footbath (t3).
Change in Distal Skin Temperature Measure (hands) from t1 to t2 | right before the footbath (t1) and right after the footbath (t2, 5-20 minutes after t1 depending on the actual footbath length)
  Distal skin temperature in °C at both hands measured with a high-definition infrared camera (FLIR-Systems, type SC660) right before (t1) and right after the footbath (t2).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, Dr., Study Director — ARCIM Institute; University of Tuebingen
Locations (1):
- Filderklinik, Filderstadt, Baden-Wurttemberg, Germany